CLINICAL TRIAL: NCT05883332
Title: A Pilot Study to Assess Effects of Self-Administered Nitrous Oxide (SANO) on Urodynamic Study (UDS) Parameters
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Heidi Rayala, Assistant Professor of Surgery, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2022P-000826
Record Dates: First submitted 2023-04-14; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: urodynamic study; nitrous oxide; neurogenic bladder; overactive bladder; ambulatory; patient experience of care
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder, Neurogenic; Urinary Bladder, Overactive | interventions — Nitrous Oxide; Oxygen

STUDY DESIGN:
Intervention Model Description: Each participant will undergo urodynamic study (UDS) with two fills. The participant will receive SANO during one fill, and oxygen during the other fill. Participants will be randomized to the order in which they receive SANO or oxygen.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participant and operating urodynamic study practitioner will be blinded to whether SANO or oxygen is given during the study fills. UDS measurements will be assessed by a blinded urologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SANO (1), Oxygen (2) (Experimental): All participants will receive self-administered nitrous oxide (SANO) at a range of 25-50% immediately before and during catheter placements. At this time, a participant-preferred level of SANO will be determined.
  At the start of the first UDS run, SANO will continue at the participant-preferred level that was determined during catheter placement, ensuring that the patient is relaxed but still conversant through the procedure.
  At the end of the first UDS run, SANO will be turned down to 0%. Participants will then receive 100% oxygen at 10 liters/minute for the duration of their second UDS run.
  Interventions: Drug: Self-Administered Nitrous Oxide; Other: Oxygen
- Oxygen (1), SANO (2) (Experimental): All participants will receive self-administered nitrous oxide (SANO) at a range of 25-50% immediately before and during catheter placements. At this time, a participant-preferred level of SANO will be determined.
  After catheter placement, SANO will be turned down to 0%. Participants will receive 100% oxygen at 10 liters/minute for the duration of their first UDS run.
  At the end of the first UDS run, SANO will start at the participant-preferred level that was determined during catheter placement, ensuring that the patient is relaxed but still conversant through the procedure. SANO will be given for the duration of their second UDS run.
  Interventions: Drug: Self-Administered Nitrous Oxide; Other: Oxygen

INTERVENTIONS:
Drug: Self-Administered Nitrous Oxide — Nitrous oxide administered at concentrations of mild sedation (20-50%)
  Other Names: nitrous oxide
Other: Oxygen — 100% oxygen at 10 Liters/minute

SUMMARY:
A urodynamic study (UDS) is a common procedure done to learn more about the cause of urinary symptoms. For some patients, UDS can be associated with anxiety or discomfort. Nitrous oxide (or laughing-gas) is a well-known sedative which is frequently used in dental offices and for pediatric procedures to reduce anxiety and pain. This study is being done to see if giving low-dose (25-50%) nitrous oxide at the time of UDS affects the measurements taken during the procedure, such as how much volume your bladder can hold, and pressures during urination. If the measurements are the same with and without self-administered nitrous oxide (SANO), it could be suggested that nitrous oxide may be a useful way of reducing patient anxiety and pain during UDS.

DETAILED DESCRIPTION:
The urodynamic study (UDS) procedure will consist of catheter placement and two "runs". Before the start of the procedure, a study staff member will assist the participant with putting on a plastic gas mask. SANO and oxygen will be given through this mask. The dose will be adjusted based on the participant's comfort level but they will not be able to request more gas than allowed. SANO will be administered during catheter placement at the start of the UDS. During the two runs, the participant will either receive SANO (run 1) then oxygen (run 2), or oxygen (run 1) then SANO (run 2).

Before the day of the UDS, participants will be asked questions related to demographics and medical history to determine study eligibility and experience of the treatment. During the UDS, participants will be asked to describe their anxiety and pain levels. Afterwards, they will be asked to complete a 15-20 minute structured interview with a study staff member to learn more about patient experience during UDS.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for urodynamic study
* Aged 21 to 85 years
* Suitable for inflation of nitrous oxide/oxygen with willingness to undergo two urodynamic study runs during the procedure
* Access to an email and computer

Exclusion Criteria:

* Perioral facial hair impeding good mask seal
* Learning disabilities and/or inability to cognitively complete survey questions
* Has any of the following medical conditions:

  1. Inner ear, bariatric or eye surgery within the last 2 weeks,
  2. Current emphysematous blebs,
  3. Severe B-12 deficiency,
  4. Bleomycin chemotherapy within the past year,
  5. Heart attack within the past year,
  6. Stroke within the past year,
  7. Class III or higher heart failure

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Bladder capacity | Measured at time of max fill during each UDS run
  Maximum liquid the bladder may hold as measured in milliliters

SECONDARY OUTCOMES:
Intra-Urodynamic Study (UDS) pain | Measured at time of max fill during each UDS run
  Pain experienced at time of max fill during each UDS run as measured by a Visual Analog Scale for Pain (VAS-P) (range: 0 [no pain] - 10 [worst pain])
Intra-Urodynamic Study (UDS) anxiety | Measured at time of max fill during each UDS run
  Anxiety experienced at time of max fill during each UDS run as measured by a Visual Analog Scale for Anxiety (VAS-A) (range: 0 [no anxiety] - 10 [worst anxiety])
Post void residual | Measured at end of void during each UDS run
  Amount of liquid left in bladder after voiding, as measured in milliliters
Max flow rate | Measured during the void at the end of each UDS run
  Maximum rate of void, as measured in milliliters per second
Detrusor overactivity | Measured during each UDS run
  Pressure sensors (which are located on the UDS catheter within the bladder) measure any bladder contractions that should not normally occur while a bladder fills. Outcome pressures will be measured in centimeters (cm) of water (H2O).
Detrusor pressure at maximum flow | Measured during each UDS run
  Pressure sensors (which are located on the UDS catheter within the bladder) measure the strength of the bladder contraction while the individual is urinating. Outcome pressures will be measured in centimeters (cm) of water (H2O).

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Rayala, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herd DW, McAnulty KA, Keene NA, Sommerville DE. Conscious sedation reduces distress in children undergoing voiding cystourethrography and does not interfere with the diagnosis of vesicoureteric reflux: a randomized controlled study. AJR Am J Roentgenol. 2006 Dec;187(6):1621-6. doi: 10.2214/AJR.05.1216. PMID 17114560

DOCUMENTS (1):
  • Informed Consent Form (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT05883332/ICF_000.pdf